CLINICAL TRIAL: NCT00318344
Title: Evaluation of Atuna Racemosa Toxicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170-06
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

INTERVENTIONS:
Drug: Atuna Racemosa

SUMMARY:
For thousands of years people in the South Pacific have used Atuna racemosa extract as a topical anti-inflammatory. We, the researchers at the Mayo Clinic, have shown this extract to also have antibacterial properties. While this extract has been used for decades in the South Pacific, a controlled clinical trial to evaluate toxicity has never been performed.

ELIGIBILITY:
The subjects will be 20 healthy male and non-pregnant, non-lactating, female volunteers of ages 18 - 65. No subject will be excluded based on minority status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Buenz, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States